CLINICAL TRIAL: NCT05923723
Title: Efficacy of a Dietary Intervention Composed of Flaxseed, Chia, and Psyllium for the Treatment of Constipation in Institutionalized Older Adults. Medellín, 2023-2024.
Brief Title: Efficacy of a Dietary Intervention for the Treatment of Constipation in Institutionalized Older Adults. Medellín, 2023-2024.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CES University (Other)
Responsible Party: Principal Investigator, Santiago Gomez Velasquez, Research Professor, doctoral student in Epidemiology and Biostatistics., CES University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Constipation psyllium
Record Dates: First submitted 2023-05-31; First posted 2023-06-28 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Constipation Chronic Idiopathic

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary intervention (Experimental)
  Interventions: Other: FIBNUTRITION
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Other: FIBNUTRITION — The dietary product selected for the study is commercially known as FIBNUTRITION, marketed in Colombia by Bio-Nutrition S.A.S with sanitary registration number NSA-001942-2016.
  Ingredients of the product:
  Flaxseed, Chia seeds, Psyllium, Polydextrose, Oat flour, Apple, Orange, Artificial flavor (Orange), Pineapple, Nopal, Xanthan gum (thickener), Silicon dioxide, Stevia (Natural sweetener), Lactobacillus Acidophilus Bifidus Casei (Prebiotics), Sodium Benzoate (Preservative), and Turmeric (Natural colorant).
  Arms: Dietary intervention
Other: Placebo — The placebo is a dietary product composed of maltodextrin, cornstarch, orange flavoring, and stevia.
  Arms: Placebo

SUMMARY:
The objective of this clinical trial is to determine if a dietary intervention for the treatment of chronic idiopathic constipation in older adults in the city of Medellin is effective (works well), focusing on the population in geriatric care centers and institutions. The goal is to obtain scientific evidence that allows determining the efficacy of this intervention for the non-pharmacological treatment of constipation in the elderly. The main question to be answered is:

"Is a dietary product designed with psyllium, chia, and flaxseed a reliable and effective treatment for managing constipation in older adults?"

The intervention and follow-up period for the study has been set at 6 weeks (45 days). During this time, participants will receive orally, once a day (every 24 hours), 1 tablespoon (20g) of the product - FIBNUTRITION - (a natural food product rich in fiber, with its main components being flaxseed, chia, and psyllium), mixed in an 8oz glass (approximately 250ml) of room temperature water using a blender (following the manufacturer's instructions for use). The product will be provided to each patient in the morning before breakfast.

The proposed research corresponds to an intervention study, specifically a randomized, controlled, double-blind, multicenter clinical trial. The researchers will compare an intervention group (dietary intervention) with a control group (placebo: a similar product that does not contain fiber or components that can alter the intestinal tract) to observe if there is a difference of at least 40% in the prevalence of satisfactory relief of constipation symptoms (desired primary effect criterion) between the two groups.

DETAILED DESCRIPTION:
Population

Older adults residing in long-term care centers in the city of Medellín who meet the diagnostic criteria of Rome IV for functional or idiopathic constipation, aged over 60 years.

Sampling Design

The sample size calculation was performed using G Power 3.1.9.7 software (78). The procedure was conducted considering a 40% difference for the desired primary outcome criterion between the two groups, assuming prevalences of 10% in the control group and 50% in the intervention group, based on previous publications with similar designs to identify a minimum clinically relevant difference (35, 79, 80). With a bilateral α of 0.05 and a statistical power of 0.8, a sample size of 46 individuals was calculated, with a 20% increase to account for potential losses or dropouts, resulting in a total of 28 individuals per group, equivalent to a final sample of 56 participants.

Estimated Start and End Dates

The start of the trial is contingent upon approval from the Doctoral Committee and the Institutional Ethics Committee of University CES. Once the research proposal is approved, the study's start date will be determined, projected for the first half of 2024. The maximum total duration of the clinical period will be two (2) months, after which the data collected will be analyzed and discussed based on the proposed analyses, followed by the presentation of results and conclusions.

Recruitment Period

This phase is projected to last a maximum of 8 weeks, with recruitment expected to begin in february 2024 and extend until june of the same year. The recruitment period will take place prior to the clinical period. The tentative deadline for accepting new cases is set for Abril 15, 2023. Prior to enrollment in the study, the principal investigator will verify compliance with inclusion criteria and the absence of exclusion criteria based on a personal interview.

Randomization Process

A block randomization procedure, also known as "permuted blocks," will be carried out to ensure periodic balance in the number of subjects assigned to each intervention group.

This procedure will be conducted in three steps:

* The size and number of blocks necessary for the study will be determined, where the size should be a multiple of the number of trial groups.
* All possible permutations within each block will be listed.
* A randomization code will be generated based on the order of selection for each block. After completing the assignments for each block, it will be verified that the same number of individuals is allocated to each group.

Intervention and Follow-up Period

The duration of intervention and follow-up for each subject in the study has been set at 6 weeks (45 days). During this time, 1 tablespoon (20g) of the product - FIBNUTRITION - will be orally administered once a day (every 24 hours) in an 8oz (approximately 250ml) glass of room temperature water, blended in a blender (following the instructions for use provided by the manufacturer). The product will be delivered to each patient in the morning before breakfast.

Adverse Events

According to the Ministry of Social Protection of Colombia, in Resolution 2378 of 2008, adverse events are defined as "any adverse medical occurrence in a patient or subject of a clinical investigation to whom a pharmaceutical product has been administered, which does not necessarily have a causal relationship with this treatment. Therefore, an adverse event (AE) can be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to it."

Additionally, the Ministry of Social Protection defines a Serious Adverse Event (SAE) as "any adverse medical occurrence in a patient or subject of a clinical investigation to whom a pharmaceutical product has been administered, which does not necessarily have a causal relationship with this treatment. Therefore, an adverse event (AE) can be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to it, which at any dose:

1. Results in death,
2. Is life-threatening,
3. Requires hospitalization of the patient or prolongation of existing hospitalization,
4. Results in persistent or significant disability/incapacity."

No serious adverse events are expected in this research due to the nature and components of the product under study. However, the possible occurrence of simple adverse events such as diarrhea, abdominal distension, or increased constipation is considered.

Recording and Reporting of Adverse Events

All adverse events that may occur during the intervention phase of the trial will be incorporated into a participant's logbook. The following steps will be followed for each adverse event:

* Due to the participants being older adults living in long-term care centers, each of these institutions has nursing staff who are aware of the research and will report any adverse events that may occur in the participants.
* In the event of an adverse event, the institution where the study is being conducted assumes responsibility for the care, assistance, and risks associated with the use of the food product.
* The report will be made to the institution's director, and if necessary, the patient's healthcare route will be activated through the social security system to which the patient is affiliated, whether it is a contributory or subsidized regime.
* The research will have the permanent availability of a gastroenterologist, who will have direct telephone communication with the nurses from each participating institution. In the event of an adverse event, the gastroenterologist will be responsible for diagnosing the severity of the event and deciding whether to activate the healthcare route.
* In the occurrence of any of the expected adverse events (diarrhea, abdominal distension, or increased constipation), the participant will be withdrawn from the study, and the treatment assignment will be suspended.
* Through the participants' characterization form (pretest), the study will establish a clear healthcare route for each participant based on their affiliation characteristics with the healthcare system (regime, healthcare provider for regular consultations, healthcare provider for emergency care).

Information Collection Techniques

Sources of Information

The study will use primary sources of information through the application of a survey designed for sociodemographic characterization and the Patient Assessment of Constipation Quality of Life Questionnaire (PAC-QOL).

Data Collection Techniques

For the identification of the study population, a characterization process will be conducted in each participating long-term care center to assess the presence of idiopathic constipation using the Rome IV criteria. Older adults who meet the clinical diagnostic criteria and the pre-defined inclusion criteria will be the study population from which the sample and respective experimental groups will be selected. The data collection process for both the intervention and control groups will be done through the completion of pretest and posttest forms, which include sociodemographic characteristics and the Patient Assessment of Constipation Quality of Life Questionnaire (PAC-QOL). The collected information will provide baseline data for the characterization of both groups to subsequently perform the respective assessment of results according to the primary and secondary criteria.

A double-blind masking process will be implemented, where neither the participants nor the investigator will know which group is assigned to the treatment. The measurement of outcomes will be conducted by the principal investigator, who will apply the respective instrument while maintaining the assigned group of each participant masked throughout the study. All participants, both in the control and intervention groups, will be assigned an alphanumeric code, and comprehensive data collection forms will be applied at each measurement point (baseline and final), ensuring privacy and autonomy in responses. Support and resolution of participants' concerns will be provided when necessary, and the complete completion of the instrument will be verified. After completing the measurements, the data will be entered into a plain Excel file.

Error and Bias Control

The study's quality control will include methodological strategies for monitoring and follow-up, aimed at improving the reliability and validity of the intervention and respective measurements.

* Selection: The strict compliance with inclusion and exclusion criteria will be directly supervised by the principal investigator. To avoid self-selection bias, the survey (Rome IV) will be described as a health survey without any mention of gastrointestinal symptoms or disorders.
* Measurement: The pretest survey will include two attention test questions with multiple-choice options, specifically asking the older adult to enter a particular response. Those who do not respond correctly to either of the questions will be excluded from the survey without completing it. The measurement methods for both clinical criteria and sociodemographic characterization of the older adult will be standardized, ensuring no measurement differences between groups. Adherence to the protocol will be supervised to ensure that the treatment was delivered to each participant as standardized. This will include protocol training and keeping a record of each delivery.
* Confounding: Variables related to pre-existing morbidities, polypharmacy, and diet will be specifically controlled. The study will focus on evaluating the group outcome in terms of satisfactory relief, rather than conducting individual analysis on each older adult.
* Matching and randomization errors: The treatment delivery will be based on a principle of simple random distribution (random assignment numbers in Excel) performed by technical personnel from the NUTRAL group. It is acknowledged that older adults with cognitive impairment may be present, resulting in difficulties in identifying symptoms or remembering their occurrence. To control this potential error, only older adults who record between 0 and 2 errors on the Pfeiffer Questionnaire (SPMSQ) to detect cognitive impairment in older adults will be included in the study.
* Intervention errors: It will be ensured that each participant receives one daily dose of the placebo or treatment in the same quantity, presentation, texture, smell, and taste to ensure masking. To avoid any contingencies where the product provider cannot continue supplying the treatment, all doses will be packaged, labeled, and properly identified for the 6-week intervention period from the start of the intervention. This means that each participant will be guaranteed the assignment of placebo or treatment for the six weeks according to the respective group. To prevent data loss from measurements, a backup will be stored in the institutional OneDrive of the University CES immediately after each data collection.
* Attrition control: The possibility of voluntary withdrawal from the study by the participating older adults is acknowledged. This attrition risk will be pre-controlled by increasing the sample size by 10% of the required value in both groups, so that the dropout of any participant does not affect the completion of the research due to missing data in the results. The principal investigator will conduct telephone follow-up with the long-term care facilities to evaluate participant retention. A face-to-face visit will be conducted in the third week to inquire about participants' satisfaction and perceptions.

Analysis Strategy

The primary analysis set will be the intention-to-treat (ITT) population, including every participant randomized with at least one post-intervention observation. In the ITT analysis, study subjects are compared within the groups they were originally assigned to, randomly. In more depth, this implies analyzing and including all patients regardless of whether they received the full treatment or withdrew or deviated from the originally established protocol. This means that patients will be analyzed as they were randomized, whether they complete the study or not (90).

Data Analysis

After preparing the database, the following analysis plan will be conducted, where variables will be addressed according to their relationship with the project's objectives, involving descriptive and analytical processing.

* Descriptive statistics will be performed based on normality tests and absolute and relative frequencies.
* Within-group comparison before and after the intervention will be conducted to determine if there are differences in the number of spontaneous evacuations. The statistical tests for this analysis will be parametric or non-parametric, depending on the distribution of the variable. The paired t-test or Wilcoxon test will be considered in this regard. Cohen's d or r-value will be used for effect size calculation for paired t-test or Wilcoxon, respectively.
* Between-group comparison at the end of the intervention will be conducted to determine if there are differences in the quality of life index. The statistical tests for this analysis will be parametric or non-parametric, depending on the distribution of the variable. The t-test or Mann-Whitney U test will be considered. Tau-b, Cliff's delta, or Cohen's d will be used for effect size calculation.
* Within-group comparison before and after the intervention will be conducted to determine if there are differences in the quality of life index. The statistical tests for this analysis will be parametric or non-parametric, depending on the distribution of the variable. The paired t-test or Wilcoxon test will be considered. Cohen's d or r-value will be used for effect size calculation for paired t-test or Wilcoxon, respectively.
* Between-group comparison at the end of the intervention will be conducted to determine if there are differences in the proportions of satisfactory relief. In this regard, the Pearson chi-square test will be considered. Phi (φ) or Cramer's V will be used for effect size calculation.

ELIGIBILITY:
Inclusion Criteria:

* Older adults aged 60 or older who meet the Rome IV criteria for functional constipation and reside in a long-term care facility in the city of Medellin (Annex 1).
* Older adults who score between 0 and 2 errors on the Pfeiffer Questionnaire (SPMSQ) to detect cognitive impairment in older adults (81). Older adults with cognitive impairment may have difficulties identifying symptoms or remembering their occurrence, which is why they will be excluded from the study

Exclusion Criteria:

* Older adults with known organic intestinal disease, a history of abdominal or pelvic radiation, previous intestinal surgery or severe liver or kidney disease, any previous abdominal or pelvic cancer, prostate problems, abdominal hernia, known intestinal cancer, and recent abdominal surgery. Other comorbidities that could interfere with the implementation or interpretation of the study.
* Older adults who have used pharmacological and non-pharmacological agents including laxatives in the two weeks prior to the start of the study will be excluded from the study.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-06-18 (Actual); Study Completion 2024-06-25 (Actual)

PRIMARY OUTCOMES:
Adequate relief at 6 weeks | 6 week
  Proportion of older adults with satisfactory relief of general constipation symptoms after 6 weeks of intervention initiation. A binary assessment measure of "satisfactory relief" (Yes/No) corresponding to the question: "In comparison to your health before starting the treatment, do you feel that the general symptoms of constipation have improved satisfactorily during the past seven days?" is used.

SECONDARY OUTCOMES:
Adequate relief at 3 weeks | 3 week
  Proportion of older adults with satisfactory relief of general constipation symptoms after 3 weeks of intervention initiation. A binary assessment measure of "satisfactory relief" (Yes/No) corresponding to the question: "In comparison to your health before starting the treatment, do you feel that the general symptoms of constipation have improved satisfactorily during the past seven days?" is used.
Change from baseline in the score of the Patient Assessment of Constipation Quality of Life (PAC-QOL). | Baseline, week 6
  Patient Assessment of Constipation Quality of Life Questionnaire (PAC-QOL). This tool consists of 28 items grouped into 4 subscales corresponding to: Concerns and Worries (11 items), Physical Discomfort (4 items), Psychosocial Discomfort (8 items), and Satisfaction (5 items). A 5-point Likert scale is used as a response scale, ranging from 0 (Not at all / Never) to 4 (Extremely / Always). A difference of 0.8 points in the overall PAC-QOL assessment (Before and after the intervention) is established as the minimally important difference (improvement) to be detected.

CONTACTS AND LOCATIONS:
Locations (2):
- Colombia (2):
  - FUNDACOL, Medellín, Antioquia
  - Prososerh, Medellín, Antioquia

IPD SHARING:
Plan to Share IPD: No